CLINICAL TRIAL: NCT07172126
Title: A Phase I/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of TQB3201 Tablets in Patients With Advanced Prostate Cancer
Brief Title: Clinical Trial to Evaluate the Tolerance of TQB3201 Tablets
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3201-I/II-01
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3201 tablets (Experimental): Each enrolled subject received 28 consecutive days of administration, once daily after meals. (25mg, 50mg, 100mg, 200mg, 400mg, 800mg, 1200mg)
  Interventions: Drug: TQB3201 tablets

INTERVENTIONS:
Drug: TQB3201 tablets — TQB3201 is an orally administered targeted protein chimera (PROTAC) drug in which one end of the drug is attached to a ligand that binds to AR and the other end to a ligand of E3 ligase (CRBN) via a linker. This product is effective against anti-androgen drugs (such as abiraterone, enzalutamide, etc.) resistance mutations, including AR amplification, point mutations (L702H, H875Y, T878A mutations, etc.), and can target the degradation of wild-type AR and AR ligand-binding domain mutants, especially L702H mutations, which is a new generation of AR-PROTAC.

SUMMARY:
TQB3201 is an orally administered targeted protein chimera (PROTAC) drug in which one end of the drug is attached to a ligand that binds to Androgen Receptor (AR) and the other end to a ligand of E3 ligase (CRBN) via a linker. The phase I phase of this trial aims to evaluate the safety, tolerability, and pharmacokinetic characteristics of TQB3201 tablets for the treatment of advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the prostate;
2. Age≥ 18 years old (calculated from the date of signing the informed consent form);
3. Eastern Cooperative Oncology Group Performance Status(ECOG )score 0-1 points;
4. Presence of metastatic disease confirmed by imaging;
5. Serum testosterone level ≤ 1.73 nmol/L (50 ng/dL) at screening;
6. Sufficient samples should be provided for gene mutation detection to determine androgen receptor gene status.
7. Patients who have progressed on the basis of at least 1 new endocrine drug;
8. The laboratory inspection meets the following standards:

   * Hemoglobin (HGB) ≥90g/L;
   * Absolute neutrophil value (NEUT) ≥1.5×109/L;
   * Platelet count (PLT) ≥75×109/L.
   * Total bilirubin (TBIL) ≤2 times the upper limit of normal (ULN); (3×ULN for patients with Gilbert syndrome ≤);
   * Alanine transferase (ALT) and aspartate transferase (AST) ≤2.5× ULN. If accompanied by liver metastasis, ALT and AST ≤ 5× ULN;
   * Serum creatinine (CR) ≤1.5× ULN or creatinine clearance estimated by the Cockcroft-Gault glomerular filtration formula ≥ 60 mL/min.
   * Urine routine: urine protein <; If the urine protein is ≥, the 24-hour urine protein quantitative ≤ 1.0 g should be confirmed.
   * Prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR) ≤1.5× ULN (no anticoagulant therapy);
   * Cardiac color ultrasound assessment: left ventricular ejection fraction (LVEF) ≥50%; > 12-lead ECG assessment: QT interval corrected by Fridericia's formula (QTcF) <450ms (males).
9. Men of childbearing potential and their partners of the opposite sex must agree to take effective contraceptive measures from the signing of the informed consent form until 6 months after the last dose of study drug;
10. Subjects voluntarily joined this study, signed the informed consent form, and had good compliance.

Exclusion Criteria:

1. Subjects with brain metastases with symptoms or symptom control time of less than 1 month;
2. Within 5 years before the first dose of medication or other malignant tumors at the same time.
3. Imaging ( Computed Tomography or Magnetic Resonance Imaging) shows that the tumor/metastasis has invaded important blood vessels, or the tumor/metastasis is very likely to invade important blood vessels during the follow-up study period, causing major bleeding;
4. Severe bone damage caused by bone metastasis; Pathological fractures and spinal cord compression of important parts that occurred within the past 6 months or are expected to occur in the near future as judged by the investigator;
5. Pleural effusion, pericardial effusion or ascites that cannot be controlled and still needs to be repeatedly drained (judged by the investigator);
6. Diseases affecting intravenous injection and intravenous blood collection, or having multiple factors affecting oral drugs (such as inability to swallow, chronic diarrhea and intestinal obstruction, etc.);
7. Adverse reactions of previous treatment have not recovered to Common Terminology Criteria (CTC) adverse event (AE) v5.0 grade ≤1, except for grade 2 alopecia, grade 2 peripheral neurotoxicity, grade 2 anemia, non-clinically significant and asymptomatic laboratory abnormalities, hypothyroidism stable on hormone replacement therapy, and other toxicities judged by the investigator to have no safety risk;
8. Have previously used or plan to use other similar drugs during the study;
9. Those who have received surgery, radiotherapy, radiotherapy, or local therapy (such as radiofrequency ablation, freezing, high-energy focused ultrasound, etc.) for prostate cancer after being diagnosed with metastatic prostate cancer;
10. Previous use of 5-ɑ reductase inhibitors within 4 weeks before the first dose; Systemic treatment with estrogens, progesterones, steroids (except for temporary use for anti-allergic use); First-generation AR antagonists; targeted therapy; biological therapy; immunotherapy; nuclide therapy; Botanicals known to have antitumor or PSA-lowering effects; Study treatments in other clinical trials.
11. Those who have undergone major surgical treatment, obvious traumatic injuries, or are allowed to undergo major surgery during the expected study treatment period within 4 weeks before the first dose, or have long-term unhealed wounds or fractures. (Major surgery is defined as: surgery of grade 3 or above in the 2022 edition of the National Surgical Grading Catalogue).
12. Subjects with any bleeding or bleeding event ≥Common Terminology Criteria for Adverse Events（CTCAE ）grade 3 within 4 weeks before the first dose.
13. Active viral hepatitis with poor control.
14. Active syphilis infection requiring treatment; Presence of active tuberculosis, history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, radiation pneumonitis requiring treatment, or active pneumonitis with clinical symptoms; Active or uncontrolled serious infection (≥CTC AE grade 2 infection);
15. Those who have a history of psychotropic substance abuse and cannot abstain from it, or have mental disorders or have a history of drug use.
16. Those who are ready to undergo or have previously received allogeneic bone marrow transplantation or solid organ transplantation, or have received hematopoietic stem cell transplantation within 60 days before the first dose, or have obvious host transplant responses;
17. Decompensated cirrhosis (Child-Pugh liver function grade B or C) or history of hepatic encephalopathy.
18. Suffering from major cardiovascular and cerebrovascular diseases；
19. Renal failure requiring hemodialysis or peritoneal dialysis;
20. History of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases;
21. Subjects who require immunosuppressive agents, or systemic, or absorbable topical hormone therapy for immunosuppressive purposes and continue to use it within 7 days prior to the first dose (daily dose of glucocorticoids <except 10 mg prednisone or other equivalent efficacy hormones);
22. Known allergy to the excipient components of the study drug;
23. History of pituitary or adrenal dysfunction;
24. Diseases that are serious or not well controlled and judged by the investigator to be at greater risk of entering this study, such as type 1 or type 2 diabetes, hyperlipidemia, thyroid disease, etc. that cannot be controlled by drugs.
25. Estimated insufficient compliance to participate in this clinical study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Up to 28days
  DLTs are defined as toxicities that occur from the first dose to the end of the first treatment cycle by the severity criteria related to the trial drug (according to Common Terminology Criteria for Adverse Events v5.0 toxicity evaluation criteria) .
Maximum tolerated dose (MTD) | Up to 28days
  The MTD was defined as the highest dose in ≥ 6 evaluable subjects without any of the following:
  1. In the DLT evaluation window, DLT occurred in 2 out of 3 subjects;
  2. In the DLT evaluation window, 1 of the first 3 subjects had DLT, and 3 more subjects were added and 1 case had ≥ DLT.
Phase II Recommended Dose (RP2D) | Up to 2 years
  The RP2D will be determined based on the safety and tolerability information of the Phase I dose escalation phase and the efficacy and safety information of the Phase II phase.
Radiographic progression-free survival (rPFS) | Up to 2 years
  The time from randomization to the first occurrence of either radiologically confirmed disease progression or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Adverse events (AEs) | Up to 2 years
  Incidence and severity of adverse events, as determined by the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grading scale.
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) and abnormal laboratory values.
The area under the curve (AUC) | cycle1 day1pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours after dose, cycle1 day7, 14 pre-dose, cycle1 day 28 pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours after dose
  The area under the curve (AUC) of serum concentration of TQB3201.
Peak concentration (Cmax) | cycle1 day1pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours after dose, cycle1 day7, 14 pre-dose, cycle1 day 28 pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours after dose
  Maximum observed concentration (Cmax) of TQB3201 antibody
Terminal half-life (T1/2) | cycle1 day1pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours after dose, cycle1 day7, 14 pre-dose, cycle1 day 28 pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours after dose
  Terminal half-life (T1/2)
Apparent Clearance (CL/F) | cycle1 day1pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours after dose, cycle1 day7, 14 pre-dose, cycle1 day 28 pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours after dose
  Apparent clearance refers to the rate of drug removal in the body, which reflects the degree of drug elimination in the body, as well as the bioavailability of the drug in the body.
Volume of Distribution at Steady State (Vss/F) | cycle1 day1pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours after dose, cycle1 day7, 14 pre-dose, cycle1 day 28 pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours after dose
  When the drug distribution in plasma and tissue reaches equilibrium, the drug distribution in the body body according to the plasma drug concentration at this time is the required body fluid volume called apparent distribution volume.
Objective Response Rate (ORR) | Up to 2 years
  Patients with soft tissue (nodes, visceral) lesions that can be evaluated according to RECIST 1.1 criteria, the proportion of cases with the best total response of soft tissue lesions as confirmed complete response (CR) and confirmed partial response (PR).
Prostate-Specific Antigen Response Rate | Up to 2 years
  Percentage of subjects whose Prostate-Specific Antigen (PSA) decreased by more than 50% from baseline and maintained for more than 4 weeks.
To PSA progression time | Up to 2 years
  Refers to the time from the start of randomization to the confirmation of PSA progression.
Time to symptomatic bone-related events (SSEs) | Up to 2 years
  Refers to the time from the randomization date to the first occurrence of symptomatic bone-related events, including the use of external beam radiation therapy (EBRT) to prevent or relieve bone symptoms, the development of new symptomatic pathological fractures (vertebral or non-vertebrae), spinal cord compression, and tumor-related orthopedic surgical intervention, whichever occurs first. Symptomatic bone-related events do not include asymptomatic fractures identified by imaging.
Overall Survival (OS) | Up to 2 years
  Refers to the time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Cancer Hospital Affiliated to Chongqing University, Chongqing, Chongqing Municipality
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Cancer Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality